CLINICAL TRIAL: NCT02236104
Title: Effect of Mechanical Insufflation-exsufflation on Respiratory Parameters in Two Neuromuscular Populations.
Acronym: coughassistAFM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: University of Versailles (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-A01042-37
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Mechanical Insufflation-exsufflation Session ( With Cough Assist)
Keywords: neuromuscular disorders; mechanical insufflation-exsufflation; respiratory parameters; plethysmography opto electronic; Vital capacity
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cough assist session (Experimental): Mechanical insufflation-exsufflation contains 15 cycles durea 2-3 seconds. pressure level fixed +/-30 cm H2O.
  Interventions: Device: Plethysmography opto electronic; Procedure: respiratory parameters

INTERVENTIONS:
Device: Plethysmography opto electronic
Procedure: respiratory parameters

SUMMARY:
A single session of Mechanical Insufflation-Exsufflation (with Cough AssistÒ) may improve airway flow and gas exchange in neuromuscular atrophy patients. The goal of this study is to confirm the beneficial effects of this treatment in a larger neuromuscular population, to study its mechanisms of action and to assess whether the effects observed persist over time. A better knowledge of this treatment should help to define its position in the respiratory management of neuromuscular patients.

DETAILED DESCRIPTION:
30 SMA and DMD adult patients will be recruited in the home ventilation unit of the intensive care department of Raymond Poincaré Hospital (Assistance Publique-Hôpitaux de Paris,Garches, France).

Respiratory parameters and comfort will be evaluated before and after (5min,

1h, 3h) a MI-E session. Vital capacity, maximal inspiratory and expiratory pressures (PImax and PEmax), peak cough flow and peak expiratory flows will be measured. Breathing pattern will be recorded allowing the measurements of respiratory frequency, tidal volume, Inspiratory time (Ti),total breath (Ttot) during tidal breathing and the calculation of tension-time index (TT0.1).

Gas exchange will be evaluated by measuring end tidal CO2, transcutaneous CO2 and pulse oxymetry.

Respiratory comfort will be assessed with a visual analog scale. Optoelectronic plethysmography will be use to perform regional ventilation evaluation. Using chest wall motion analysis we will compute respiratory participation of upper, lower thorax and abdomen, right and left side.

Results should allow to analyse the effects of MI-E on regional ventilation. The mechanisms of action of MI-E on respiration and chest-wall motion will be analysed and the persistence of the beneficial effect of MI-E will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged more than 18 years
* Written consents
* Neuromuscular disorders
* Hemodynamic stability

Exclusion Criteria:

* Pulmonary disorder
* Acute respiratory failure
* Cognitive deficit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
maximal inspiratory pressures | 2 hours
  measure of maximal inspiratory pressures before mechanical insufflation-exsufflation session, just after this session and an hour after.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic LOFASO, MD PHD, Principal Investigator — Raymond poincare hospital; Michel Petitjean, MDPHD, Principal Investigator — Raymond Poincare hospital
Locations (1):
- Hopital Raymond Poincaré, Garches, Garches, France